CLINICAL TRIAL: NCT07231692
Title: Comparative Evaluation of Biceps Femoris Short Head (BiFeS) and Adductor Canal Block and Interspace Between the Popliteal Artery and Capsule of the Knee (IPACK) and Adductor Canal Block Combinations for Postoperative Pain After Total Knee Arthroplasty
Brief Title: Comparison of BiFeS + ACB and IPACK + ACB Block Combinations for Postoperative Pain After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Elif Sarikaya Ozel, Anesthesiologist, Principal Investigator, Karabuk University
Other Study IDs: BiFeS2025/2462
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pain After Total Knee Arthroplasty; Pain, Postoperative; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group BiFeS: Adductor canal block and BiFeS block ( 15 ml %0.25 bupivacaine and 25 ml %0.25 bupivacaine) + IV morphine patient-controlled analgesia (PCA)
- Group IPACK: Adductor canal block and IPACK block ( 15 ml %0.25 bupivacaine and 25 ml %0.25 bupivacaine) + IV morphine patient-controlled analgesia (PCA)

SUMMARY:
This prospective observational study will compare the postoperative analgesic efficacy of two multimodal regional anesthesia combinations routinely used after total knee arthroplasty (TKA) performed under spinal anesthesia. The study will observe patient groups who receive, as part of standard clinical practice, either the Biceps Femoris Short Head (BiFeS) block combined with the Adductor Canal Block (ACB) or the Interspace Between the Popliteal Artery and the Capsule of the Knee (IPACK) block combined with the Adductor Canal Block (ACB). The research team will not assign, perform, or direct any blocks; all regional anesthesia procedures will be administered independently by anesthesiologists experienced in ultrasound-guided regional anesthesia as part of routine care.

Postoperative pain will be observed and documented using the Numeric Rating Scale (NRS) at multiple time points within the first 24 hours. Opioid consumption will be recorded based on intravenous patient-controlled analgesia (PCA) data, and the need for rescue analgesia will be noted. Additional postoperative observations will include functional recovery, quality of recovery scores, and the incidence of adverse events.

Postoperative pain will be evaluated using the Numeric Rating Scale (NRS) at multiple time points within the first 24 hours. Opioid consumption will be recorded through intravenous patient-controlled analgesia (PCA), and the need for rescue analgesia will be assessed. Additional postoperative observations will include functional recovery, quality of recovery scores, and the incidence of adverse events.

DETAILED DESCRIPTION:
This prospective, single-center, observational study will be conducted at Karabük Training and Research Hospital. This is an observational study. Participants are not assigned to any intervention by the research team. All regional anesthesia blocks are performed as part of routine clinical practice, and the investigators only collect data related to outcomes. No interventions are administered because of study participation. The research team does not perform, modify, or direct any clinical procedures; all blocks are performed independently as part of routine care.

The study population will include adults aged 18-80 years undergoing elective unilateral total knee arthroplasty (TKA) under spinal anesthesia. All eligible patients will receive routine multimodal analgesia and will undergo one of two commonly used regional anesthesia combinations:

Biceps Femoris Short Head (BiFeS) block + Adductor Canal Block (ACB)

Interspace Between the Popliteal Artery and the Capsule of the Knee (IPACK) block + Adductor Canal Block (ACB)

The choice of block combination will be determined by the attending anesthesiologist as part of standard clinical practice. The research team will not influence clinical decisions and will only record perioperative and postoperative data.

Regional Anesthesia Techniques (Routine Care Descriptions)

IPACK Block: The patient will remain in the supine position with the knee flexed 30-45°. A 3.5-6 MHz convex US probe will be placed over the popliteal fossa to visualize the popliteal artery at the femoral condyle level in the short axis. A 22G, 100 mm needle will be advanced in-plane from lateral to medial, and the tip will be positioned between the popliteal artery and femoral condyle. After negative aspiration, 25 mL 0.25% bupivacaine will be slowly injected.The aim is to provide effective posterior knee analgesia by blocking the sensory branches without motor impairment.

BiFeS Block: With the patient in the supine position, the potential space between the lateral supracondylar line of the femur and the short head of the BF muscle will be identified under US guidance. A 22G, 100 mm echogenic needle will be advanced in-plane, and 25 mL 0.25% bupivacaine will be injected. All blocks will be performed by anesthesiologists experienced in ultrasound-guided regional anesthesia.

ACB: ACB will also be performed in the same session using 15 mL 0.25% bupivacaine beneath the sartorius muscle under US guidance.

Anesthesia and Analgesia Approach

All patients will undergo spinal anesthesia as part of routine care. Postoperative analgesia will include multimodal medications used in standard practice at the study center, as well as intravenous patient-controlled analgesia (PCA) when required. Pain intensity will be assessed using the Numeric Rating Scale (NRS), an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Opioid use will be calculated in morphine milligram equivalents (MME).

Outcome Assessments

Postoperative outcomes will include cumulative opioid consumption at 12 and 24 hours, pain scores at predefined time points, quality of recovery using the Quality of Recovery-15 (QoR-15) questionnaire, postoperative nausea and vomiting (PONV) scores, block performance time, time to first mobilization, functional evaluation with the Timed Up and Go (TUG) test, block-related and opioid-related complications, and total length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years scheduled for elective unilateral total knee arthroplasty (TKA) under spinal anesthesia
* ASA physical status I-III
* Eligible for and capable of using patient-controlled analgesia (PCA)
* Provided written informed consent

Exclusion Criteria:

* Chronic opioid use for more than four weeks before surgery
* Presence of chronic pain conditions (e.g., migraine, fibromyalgia)
* History of alcohol or drug abuse
* Known allergy or hypersensitivity to local anesthetics or opioids
* Severe organ dysfunction (e.g., significant hepatic or renal disease)
* Revision or bilateral knee arthroplasty
* Contraindications to regional anesthesia
* Preexisting neuropathy or prior femoral vascular surgery on the operated side.
* Infection near the injection site (e.g., osteomyelitis, septic joint).
* Contraindication to spinal anesthesia (e.g., refusal, coagulopathy, use of anticoagulants or antiplatelet agents) or inability to understand NRS.
* Severe psychiatric or cognitive disorders (e.g., psychosis, dementia) that prevent cooperation or pain assessment
* Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients aged 18-80 years undergoing elective unilateral total knee arthroplasty (TKA) under spinal anesthesia at Karabük Training and Research Hospital. Eligible participants will have ASA physical status I-III and be capable of using patient-controlled analgesia (PCA). Patients will be prospectively observed as part of routine multimodal analgesia including either BiFeS + ACB or IPACK + ACB block combinations for postoperative pain management.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours after surgery will be measured. Patients will be able to request opioids via a PCA device when their NRS score is ≥ 4.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 12 hours after surgery | postoperative 12th hour
  Morphine consumption in the first 12 hours after surgery will be measured. Patients will be able to request opioids via a PCA device when their NRS score is ≥ 4.
Postoperative pain scores | Postoperative day 1
  Pain status at rest and while activity will be assessed by numeric rating scale (NRS) score at 0, 3, 6, 12, 18 and 24 hours after surgery. In addition, the time until the first analgesic requirement will be recorded. The NRS is an 11-point numeric scale that ranges from 0 to 10.
Block performance time | İntraoperative period
  The duration of block performance will be recorded for BiFeS, ACB, and IPACK procedures. Time will be measured in seconds from the placement of the ultrasound probe on the skin to the completion of local anesthetic injection.
The Quality of Recovery-15 (QoR-15) score | 24 hours postoperatively and postoperative day 2-4
  Patient recovery quality and satisfaction will be assessed using the QoR-15 questionnaire at 24 hours postoperatively and at discharge. Higher scores indicate better recovery (QoR-15 score [0-150]).
The postoperative nausea and vomiting (PONV) scores and the number of patients requiring antiemetic medication | Postoperative day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18 and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required (The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once).
Time of first analgesic request | Postoperative day 1
  Time at which the first analgesic is requested
Number of patients requiring rescue analgesia | Postoperative day 1
  Number of patients who required additional rescue analgesics (IV tramadol 100 mg) despite PCA use will be recorded.
Block-related complications | Postoperative day 7
  Complications related to the block procedure, such as local bleeding, hematoma, infection, or local anesthetic systemic toxicity (LAST), will be recorded.
Opioid-related side effects | Postoperative day 7
  Adverse effects including pruritus, sedation, fatigue, or respiratory depression associated with opioid use will be documented.
Timed Up and Go (TUG) test duration | Postoperative day 1
  The time (in seconds) taken for the patient to rise from a chair, walk 3 meters, return, and sit down will be recorded as a measure of functional mobility.
Time to first mobilization | Postoperative day 1 and postoperative day 2-4
  Time elapsed from the end of surgery to the patient's first mobilization (standing and walking with physiotherapist assistance) will be recorded.
Length of hospital stay | From surgery to postoperative day 2-4
  Total time from entry to the operating room until discharge from the hospital will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Sarikaya Özel, M.D., Principal Investigator — Karabuk Training and Research Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Karabuk Training and Research Hospital, Department of Anesthesiology and Reanimation, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No